CLINICAL TRIAL: NCT04021901
Title: A Prospective Multicenter Study of Balloon Dilatation for the Treatment of Benign
Brief Title: A Study of Balloon Dilatation for the Treatment of Benign Ureteral Stricture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Yinghao Sun, Director of Urology department, Changhai Hospital
Other Study IDs: SHOT-20181112
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Stricture Ureter
Keywords: benign ureteral stricture; balloon dilatation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- F21: balloon diameter F21
  Interventions: Device: balloon dilatation
- F24: balloon diameter F24
  Interventions: Device: balloon dilatation

INTERVENTIONS:
Device: balloon dilatation — The balloon catheter (BD U30) was placed through narrow ureter along the guide wire, and the balloon was pressurized to 25 atm until the "bee waist sign" disappeared on the balloon or the narrow section was seen under the endoscope. Dilation, expansion for 10 min, and then through the endoscope to observe the stenosis of the stenosis (stenosis of the stenosis of the visible adipose tissue)

SUMMARY:
This study is designed to treat benign ureteral stricture with balloon dilatation through prospective multicenter studies. It aims to indications, procedure standards, and therapeutic effects of balloon dilation, and provide further guidance for endoscopic treatment of benign ureteral stricture.

DETAILED DESCRIPTION:
Benign ureteral stricture refers to a urinary tract obstruction caused by a partial or full ureteral lumen that is less normal than normal. It can lead to urinary dilatation, water accumulation, and renal colic in the upper segment of the stenosis. If treat not in time, it will affect renal function and even causes irreversible kidney failure.In recent years, with the development of endoscopic techniques, it provides a cost-effective and less invasive treatment for the treatment of ureteral stricture. In recent years, with the development of endoscopic techniques, it has provided a cost-effective and less invasive treatment for the treatment of ureteral stricture, and has achieved satisfactory results. Therefore, more and more urologists choose to treat ureteral stricture under endoscopy. The techniques of urinary endoscopic treatment of benign ureteral stricture include ureteral balloon dilatation, ureteral holmium laser incision, and ureteral stent implantation. Among them, the ureteral balloon dilatation technique is characterized by the use of a balloon to uniformly force the ureteral wall, tearing the narrow scar tissue, expanding the inner diameter of the ureter, recanalizing the urinary tract, and alleviating hydronephrosis. It have been reported with less complications and simple procedure. However, there's still no consensus on its treatment indication，procedure standards and curative effect. This study is designed to treat benign ureteral stricture with balloon dilatation through prospective multicenter studies. It aims to indications, procedure standards, and therapeutic effects of balloon dilation, and provide further guidance for endoscopic treatment of benign ureteral stricture.

ELIGIBILITY:
Inclusion Criteria:

* • Subject has provided informed consent and indicated a willingness to comply with study treatments

  * Subject is 18-70 yrs of age
  * Subject can be either male or female
  * Subject diagnosed with ureteral stricture or atresia by enhanced CTU, intravenous pyelography or retrograde pyelography;
  * Subject's ureteral stenosis length is ≤ 2cm (single or multiple segments)

Exclusion Criteria:

* • Subject has any congenital ureteral anatomical deformity, abdominal organ compression, oppression caused by malignant tumor metastasis

  * Subject has poor result after endoscopic balloon dilatation treatment
  * Subject has a GFR <25% on the affected side of the kidney
  * Subject has an active urinary tract infection (e.g., cystitis, prostatitis, urethritis, etc.)
  * Subject has been diagnosed with a urethral stricture or bladder neck contracture
  * Subject has been diagnosed with a urinary tract infection related to stone obstruction within two weeks
  * Subject has severe hematuria that might blur the vision of the endoscopy
  * Subject is pregnant or in monthly period
  * Subject has coexistent disease like systemic disease, heart disease, lung disfuction or other diseases that could not tolerate the endoscopic surgery or anesthesia.
  * Subject has unadjusted diabetes or high blood pressure
  * Subject has a disorder of the coagulation cascade system that would put the subject at risk for intraoperative or postoperative bleeding
  * Subject is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (2 weeks)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ureteral stricture or atresia by enhanced CTU, intravenous pyelography or retrograde pyelography, and ureteral stenosis length is ≤ 2cm (single or multiple segments)
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment success in follow-up results after 6 months | 6 months after surgery
  The treatment is effective (satisfying any of the following 3 items, that is, the treatment is considered effective) Treatment failure (not satisfying any of the following 3 items is invalid, that is, treatment failure)
  1. Retrograde pyelography normal development;
  2. ECT shows improvement in renal function on the affected side;
  3. CT shows the reduced hydronephrosis.

SECONDARY OUTCOMES:
Rate of treatment success during the operation | Intraoperative
  1. Effective: the balloon is expanded through the stenosis segment, and the diameter of the ureteral tube is obviously thickened after expansion, and the scar tissue is obviously torn, and the surrounding adipose tissue is visible;
  2. Failure: The guidewire or balloon cannot pass through the stenotic segment of the ureter and cannot expand the stenosis (the scar tissue is not torn).

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong H, Peng Y, Li L, Gao X. Prevention strategies for ureteral stricture following ureteroscopic lithotripsy. Asian J Urol. 2018 Apr;5(2):94-100. doi: 10.1016/j.ajur.2017.09.002. Epub 2017 Sep 22. PMID 29736371
- [Background] Lojanapiwat B, Soonthonpun S, Wudhikarn S. Endoscopic treatment of benign ureteral strictures. Asian J Surg. 2002 Apr;25(2):130-3. doi: 10.1016/S1015-9584(09)60160-3. PMID 12376232
- [Background] Kramolowsky EV, Tucker RD, Nelson CM. Management of benign ureteral structures: open surgical repair or endoscopic dilation? J Urol. 1989 Feb;141(2):285-6. doi: 10.1016/s0022-5347(17)40742-7. PMID 2913345
- [Background] Fasihuddin Q, Abel F, Hasan AT, Shimali M. Effectiveness of endoscopic and open surgical management in benign ureteral strictures. J Pak Med Assoc. 2001 Oct;51(10):351-3. PMID 11768936
- [Background] Brooks JD, Kavoussi LR, Preminger GM, Schuessler WW, Moore RG. Comparison of open and endourologic approaches to the obstructed ureteropelvic junction. Urology. 1995 Dec;46(6):791-5. doi: 10.1016/S0090-4295(99)80345-8. PMID 7502417
- [Background] Chandhoke PS, Clayman RV, Stone AM, McDougall EM, Buelna T, Hilal N, Chang M, Stegwell MJ. Endopyelotomy and endoureterotomy with the acucise ureteral cutting balloon device: preliminary experience. J Endourol. 1993 Feb;7(1):45-51. doi: 10.1089/end.1993.7.45. PMID 8481721
- [Background] Bromwich E, Coles S, Atchley J, Fairley I, Brown JL, Keoghane SR. A 4-year review of balloon dilation of ureteral strictures in renal allografts. J Endourol. 2006 Dec;20(12):1060-1. doi: 10.1089/end.2006.20.1060. PMID 17206902
- [Background] Liu JS, Hrebinko RL. The use of 2 ipsilateral ureteral stents for relief of ureteral obstruction from extrinsic compression. J Urol. 1998 Jan;159(1):179-81. doi: 10.1016/s0022-5347(01)64050-3. PMID 9400466
- [Background] Ravery V, de la Taille A, Hoffmann P, Moulinier F, Hermieu JF, Delmas V, Boccon-Gibod L. Balloon catheter dilatation in the treatment of ureteral and ureteroenteric stricture. J Endourol. 1998 Aug;12(4):335-40. doi: 10.1089/end.1998.12.335. PMID 9726399
- [Result] Tyritzis SI, Wiklund NP. Ureteral strictures revisited...trying to see the light at the end of the tunnel: a comprehensive review. J Endourol. 2015 Feb;29(2):124-36. doi: 10.1089/end.2014.0522. Epub 2014 Oct 23. PMID 25100183